CLINICAL TRIAL: NCT06753006
Title: A Study of Neurorehabilitation Based on Robotics, Brain-Computer Interface (BCI) and Virtual Reality (VR) in Patients with Upper Limb Paresis Due to Stroke in the Early Rehabilitation Period
Brief Title: Research on the Effectiveness of Neurorehabilitation After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurotechnika (Industry)
Collaborators: Samara State Medical University (Other); Samara Regional Clinical Hospital V.D. Seredavin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NT-STROKE-2024-09
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Stroke Acute; Stroke with Hemiparesis; Stroke, Acute; Stroke, Acute, Ischemic; Stroke, Ischemic
Keywords: Stroke; Rehabilitation; Brain-Computer Interface; Motor Imagery; Robotics; Virtual Reality; Neurofeedback
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either one of three experimental groups or a control group.
Who Masked: Outcomes Assessor
Masking Description: Participants will be evaluated by blinded assessors before being assigned to one of the study arms, and their rehabilitation outcomes will also be assessed by blinded assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (4):
- Control (Active Comparator): The Control group receives a standard course of intervention (14-21 days) as prescribed by the attending physician, in accordance with the standards of the Ministry of Health of the Russian Federation for the provision of medical care to people who have suffered a stroke.
  Interventions: Procedure: Standard course
- MI+VR (Experimental): In addition to the standard course of intervention, the MI+VR group undergoes 10-12 sessions using a novel simulator involving the paretic arm with immersion in virtual reality.
  Interventions: Device: Neurorehabilitation simulator; Procedure: Standard course
- MI2+VR (Experimental): In addition to the standard course of intervention, the MI2+VR group undergoes 10-12 sessions using a novel simulator involving both arms (healthy and paretic) with immersion in virtual reality.
  Interventions: Device: Neurorehabilitation simulator; Procedure: Standard course
- MI2 (Experimental): In addition to the standard course of intervention, the group MI2 undergoes 10-12 sessions using a novel simulator involving both arms (healthy and paretic) without immersion in virtual reality, using a computer display instead.
  Interventions: Device: Neurorehabilitation simulator; Procedure: Standard course

INTERVENTIONS:
Device: Neurorehabilitation simulator — The participant must complete a mental task - imagine the movement of his arm. If successful, the robotic simulator moves the paralyzed limb.
  Arms: MI+VR; MI2; MI2+VR
Procedure: Standard course — The participant receives a standard course of intervention as prescribed by the attending physician in accordance

SUMMARY:
This clinical trial aims to investigate the effectiveness of a novel neurorehabilitation technology for treating stroke in adults. The study will evaluate a simulator that combines robotic orthosis, a non-invasive brain-computer interface (BCI), and a virtual reality (VR) display. The goal of this trial is to advance stroke rehabilitation by exploring the potential benefits of these cutting-edge technologies.

Key Research Questions:

Efficacy: Does the new simulator significantly improve arm function compared to standard rehabilitation techniques?

BCI Technology: Which approach - motor imagery of only the paretic arm or both the paretic and healthy arm - yields greater functional improvements?

VR Contribution: How does the integration of VR enhance rehabilitation outcomes?

Safety and Tolerability: What potential side effects or adverse events may arise from using the new simulator?

Participants who have suffered a stroke will undergo a standard rehabilitation course, during which 10-12 sessions will take place using the innovative simulator: a robotic device moves a patient's paralyzed arm at the command of a non-invasive brain-computer interface to perform a game task resembling real-life activities, augmented by a virtual reality display.

Researchers will assess the impact of the new technology on arm function to determine its efficacy in promoting recovery.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age 18 to 80 years at the time of stroke onset.
* Early rehabilitation period (up to 6 months post-stroke).
* Diagnosis of acute cerebrovascular accident confirmed by MRI or CT.
* Upper limb paresis severity between 0 and 3 on the 6-point Medical Research Council (MRC) muscle strength scale.
* Ability and willingness to comply with the study protocol.
* Demonstrated motivation for rehabilitation.

Exclusion Criteria:

* Montreal Cognitive Assessment scale (MoCA) score less than 10 points.
* Hamilton Depression Rating Scale (Ham-D) score greater than 18 points.
* Modified Rankin Scale (mRS) score greater than 4 points.
* Pre-existing conditions that cause decreased muscle strength or increased muscle tone in the upper limbs (e.g., cerebral palsy, traumatic brain injury) or rigidity (e.g., Parkinson's disease, contractures).
* Advanced arthritis or significant limitation of upper limb range of motion.
* Absence of part of the upper limb due to amputation for any reason.
* Any medical condition that may affect the conduct of the study or patient safety (e.g., mental illness).
* Alcohol abuse or recreational drug use within the 12 months preceding the study.
* Use of experimental medications or medical devices within the 30 days preceding the study.
* Inability to comply with research procedures, as determined by the researcher.
* The severity of the patient's condition, based on neurological or physical status, does not permit full rehabilitation.
* Visual acuity less than 0.2 in the weakest eye according to the Sivtsev visual acuity chart.
* Unstable angina and/or heart attack within the 30 days preceding the study.
* Recurrent stroke.
* Uncontrolled arterial hypertension.
* Ataxia.
* Presence of a pacemaker and/or other implanted electronic devices.
* Use of muscle relaxants.
* Peripheral neuropathy.
* Coexisting diseases in an exacerbation or decompensated stage requiring active treatment.
* Allergic reactions or other skin lesions at the EEG electrode application sites at the time of the study.
* Acute urinary tract infections.
* Acute thrombophlebitis.
* Any form of epilepsy.
* Benign and malignant neoplasms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
FMA-UE A-D | From enrollment to the end of treatment at 2-3 weeks
  The Fugl-Meyer Assessment for Upper Extremity, parts A-D (FMA-UE A-D) evaluates a patient's motor function, with scores ranging from 0 (indicating the most severe impairment) to 66 (indicating no impairment). Details available at https://www.gu.se/en/neuroscience-physiology/fugl-meyer-assessment.
ARAT | From enrollment to the end of treatment at 2-3 weeks
  The Action Research Arm Test (ARAT) evaluates a patient's ability to handle objects of various sizes, weights, and shapes, making it a specific measure of arm-related activity limitations. Scores range from 0 (indicating the most severe impairment) to 57 (indicating no impairment). Details available at https://strokengine.ca/en/assessments/action-research-arm-test-arat.

SECONDARY OUTCOMES:
NIHSS | From enrollment to the end of treatment at 2-3 weeks
  Dynamics according to the National Institutes of Health Stroke Scale (NIHSS) that assesses a stroke patient's neurological impairment and degree of recovery for patients with stroke in the range from 0 (no impairment) to 42 (very severe impairment). Details available at https://strokengine.ca/en/assessments/nihss.
Ashworth | From enrollment to the end of treatment at 2-3 weeks
  Dynamics according to the Ashworth Spasticity Scale that assesses a patient's spasticity in the range from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). Details available at https://www.sralab.org/rehabilitation-measures/ashworth-scale-modified-ashworth-scale.
RMI | From enrollment to the end of treatment at 2-3 weeks
  Dynamics according to the Rivermead Mobility Index (RMI) that assesses a patient's functional abilities such as gait, balance, and transfers in the range from 0 (worst mobility performance) to 15 (best mobility performance). Details available at https://strokengine.ca/en/assessments/rivermead-mobility-index-rmi.
MRS | From enrollment to the end of treatment at 2-3 weeks
  Dynamics according to the Modified Rankin Scale (MRS) that assesses a patient's level of functional independence in the range from 0 (no symptoms) to 5 (severe disability). Details available at https://strokengine.ca/en/assessments/modified-rankin-scale-mrs.
SF-36 | From enrollment to the end of treatment at 2-3 weeks
  The SF-36 is a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being. Scores range from 0 (maximum disability) to 100 (no disability). Details available at https://nexusipe.org/advancing/assessment-evaluation/short-form-sf-36-health-survey.

OTHER OUTCOMES:
ICF | From enrollment to the end of treatment at 2-3 weeks
  The International Classification of Functioning, Disability and Health, known more commonly as ICF, is a classification of health and health-related domains. The ICF will be used to assess the impairment of body functions resulting from a stroke. Details available at https://www.who.int/standards/classifications/international-classification-of-functioning-disability-and-health

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zakharov, Ph.D., Principal Investigator — Samara State Medical University
Locations (1):
- Samara Regional Clinical Hospital named after V.D. Seredavin, Samara, Samara Oblast, Russia

IPD SHARING:
Plan to Share IPD: No
Only authorized members of the research team will have access to individual participant data (IPD). The research team will not share any IPD with third parties. However, de-identified demographic and clinical data-such as treatment details, baseline characteristics, and outcome measures-will be made publicly available.